CLINICAL TRIAL: NCT02373228
Title: Optimization of Music Compression for People With Hearing Impairment
Brief Title: Optimization of Music Compression
Acronym: OMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Phonak AG, Switzerland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: KEK-ZH 2014-0520
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Compressive signal processing algorithm (Experimental): Participants compare music signals with preprocessing to the same music signals without compressive preprocessing.
  Interventions: Other: Audio signal processing (applied offline before playback)

INTERVENTIONS:
Other: Audio signal processing (applied offline before playback)

SUMMARY:
Hearing impaired persons suffer from inferior music perception with and without hearing aids. Hearing aids, however, are primarily designed to improve speech intelligibility not music enjoyment. This study investigates the potential benefit of signal processing strategies that are optimized for music. The purpose of this study is to improve music compression for hearing impaired people.

ELIGIBILITY:
Inclusion Criteria:

* Female and male adults between 18 and 99 years
* German-speaking
* Symmetric, mild to severe, ski-slope hearing loss
* Binaural hearing aid user without frequency lowering
* Informed Consent as documented by signature

Exclusion Criteria:

* Have taken part in a study at Phonak within 4 months prior to the first session
* People with mental-health problems
* People whose audiogram is older than 12 months and it is not possible make a reliable measurement
* Very limited motor activity or mobility

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Benefit of signal processing for music perception | 3 months
  Participants rate the enjoyment of music in 4 separate sessions, spread over an anticipated time frame of 3 months.

SECONDARY OUTCOMES:
Performance in music discrimination tests | 3 months
  Participants perform an adaptive music discrimination test in which their discrimination thresholds are measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Phonak AG, Staefa, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Kirchberger M, Russo FA. Dynamic Range Across Music Genres and the Perception of Dynamic Compression in Hearing-Impaired Listeners. Trends Hear. 2016 Feb 10;20:2331216516630549. doi: 10.1177/2331216516630549. PMID 26868955